CLINICAL TRIAL: NCT06872112
Title: Phase I Study: A Dose-Escalation Study Evaluating the Safety and Tolerability of Artesunate in Patients With Pulmonary Arterial Hypertension
Brief Title: A Study Evaluating the Safety and Tolerability of Artesunate in Patients With Pulmonary Arterial Hypertension
Acronym: (STOP-PAH)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph C. Wu (Other)
Responsible Party: Sponsor-Investigator, Joseph C. Wu, Director, Stanford Cardiovascular Institute, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 80578
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: Pulmonary Arterial Hypertension; Artesunate; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Treatment Arm (Experimental): Dose escalating study with a Follow-up (washout) Period:
  Total study period of the open-label study: 14 weeks Screening Period: up to 4 weeks Treatment Period (20 mg TID): 4 weeks Treatment Period (40 mg TID): 4 weeks Treatment Period (60 mg TID): 4 weeks Follow-up (washout) Period: 2 weeks after treatment period ends
  Interventions: Drug: Artesunate

INTERVENTIONS:
Drug: Artesunate — Participants will receive artesunate capsules. Participants will receive artesunate capsules TID in a dose escalation manner (60 mg, 120 mg, 180 mg total daily).

SUMMARY:
This is a 20-week, Phase 1, single-center, open-label, dose-escalation study evaluating the safety and tolerability of daily oral artesunate in patients with PAH.

ELIGIBILITY:
Inclusion Criteria

* Each participant must meet the following criteria to be enrolled in this study:
* Adults aged 18 to 75 years.
* WHO functional class I, II/III despite treatment with maximally tolerated doses of 2 or more treatment modalities including PDE5 inhibitors, guanylate cyclase stimulators, endothelin receptor antagonists, and prostanoids when appropriate.

Exclusion Criteria

* Participants who meet any of the following criteria will be excluded from the study.
* Participants with serious concomitant morbidity per investigator assessment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with treatment-related Adverse Events (AEs) and Serious Adverse Events (SAEs) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roham Zamanian, MD, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No